CLINICAL TRIAL: NCT02154568
Title: Flow Quantification in the Human Airways Using Hyperpolarized Helium 3 MRI
Brief Title: Study of Airflow in the Lungs Using Helium MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16885; W81XWH-09-2-0027 (Other Grant/Funding Number: US Army Medical Research Acquisition Activity)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: COPD; Healthy; Constrictive Bronchitis
Keywords: Hyperpolarized gas MRI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperpolarized helium MRI of the chest (Experimental)
  Interventions: Drug: hyperpolarized helium MRI of the chest

INTERVENTIONS:
Drug: hyperpolarized helium MRI of the chest — Using hyperpolarized helium as an inhaled gaseous contrast agent for MRI, we will measure the velocity of inhaled breath in the trachea.

SUMMARY:
Computer simulations are being developed to predict air flow abnormalities in the airways of patients with lung disease. The purpose of this study is to obtain actual gas flow measurements in the lungs of healthy patients and patients with lung disease and use these measurements to validate the computer models.

DETAILED DESCRIPTION:
The Biotechnology High Performance Computing Software Applications Institute (BHSAI) of the Department of Defense (DoD) is studying airflow in the lungs using computational fluid dynamics in order to characterize disease-specific airflow patterns and provide useful information for medical applications. To validate these models, they are seeking to obtain experimental data of airflow in human lungs, both healthy and diseased. An assessment of airflow can be obtained by using hyperpolarized noble gas (HNG) magnetic resonance imaging (MRI) or, more specifically, hyperpolarized helium-3 (HHe) MRI in conjunction with flow-encoding schemes that are well-established in conventional proton MRI

Four chronic obstructive pulmonary disease (COPD) patients and four healthy subjects will undergo pulmonary function tests (PFTs), computed tomography (CT) scan covering the mouth, neck, and chest, and hyperpolarized helium 3 MRI. Before and after the MRI scans, three spirometry readings will be taken while the subject is lying in the same position as in the MR scanners. Data will be analyzed by the BHSAI. UVa will provide the de-identified raw image data and the de-identified results of the spirometry and other tests to BHSAI

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects:

  * Normal PFT values: FEV1 > 90% predicted; and Forced vital capacity (FVC) > 90% predicted
  * Normal chest x-ray (CXR)
  * Medical history: No active pulmonary symptoms (cough, shortness of breath, sputum); Negative history of pulmonary disease; Negative smoking history (never smoked)
* Pulmonary Disease Subjects:

  * PFT values: FEV1/FVC < 70% (indicative of obstruction); and 30% < FEV1 < 50% predicted
  * CXR normal except hyperinflation
  * Symptoms - chronic shortness of breath
* All test subjects, healthy and with COPD should have similar physical anthropometric characteristics:

  * Similar age with age difference less than 3 years
  * Similar height (within 3-4 inches)

Exclusion Criteria:

* Any condition for which a MRI procedure is contraindicated.
* Presence of any non-MRI compatible metallic material in the body, such as pacemakers, metallic clips, etc.
* Likelihood of claustrophobia
* Chest circumference greater than that of the helium MR coil.
* Pregnancy, by report of subject. Clinically in the Department of radiology at UVA, self report is used when screening patients for MR scans as well as CT scans and fluoroscopy studies. If the subject reports there is any chance of their being pregnant a urine pregnancy test will be performed prior to any imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-11; Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Hyperpolarized helium MRI flow velocity map | Day 1
  Using hyperpolarized helium as an inhaled contrast agent for MRI, we will measure the velocity of inhaled breath in the trachea.

SECONDARY OUTCOMES:
Hyperpolarized helium MRI flow velocity map | Day1
  Spirometry (FEV1)
Hyperpolarized helium MRI flow velocity map | Day 1
  Spirometry (FVC)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States